CLINICAL TRIAL: NCT06354153
Title: Influence of Polarity Management Training Program on First Line Nurse Manager Creativity Behavior and Motivation
Brief Title: Polarity Management Training Program for First Line Nurse Manager
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Nagah Abd El-Fattah Mohamed Aly, Assistant professor of Nursing administration, Matrouh University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0305898
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Intervention; Knowledge, Attitudes, Practice
Keywords: Polarity; Management; Training Program; Nurse Managers; Creativity; Motivation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: A quasi-experimental design utilized one group for pre-, post, and follow-up intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group of first-line nurse managers (Other): First-line nurse managers received a polarity training program
  Interventions: Other: Polarity Management Training Program
- intervention group (Other): 60 first-line nurse managers received a polarity training program
  Interventions: Other: Polarity Management Training Program

INTERVENTIONS:
Other: Polarity Management Training Program — 60 first-line nurse managers received a training program involving theoretical and practical sessions

SUMMARY:
Polarities are vital issues in healthcare systems. Nursing is a profession riddled with polarities. If first-line nurse managers are well trained to manage polarities in the workplace, this could lead to positive outcomes for nurses, nurse managers and organization performance.

DETAILED DESCRIPTION:
Polarities are vital issues in healthcare systems. Nursing is a profession riddled with polarities. If first-line nurse managers are well trained to manage polarities in the workplace, this could lead to positive outcomes for nurses, nurse managers and organization performance. This study aimed to examine the influence of polarity management training program on first-line nurse managers' creative behavior and motivation.

ELIGIBILITY:
Inclusion Criteria:

First-line nurse managers

* willing to participate in the study
* work in all inpatient care units of Alexandria University hospitals
* Sign a consent

Exclusion Criteria:

First-line nurse managers

* work in outpatient units
* Did not sign a consent
* Absent from training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure nurse managers' knowledge | one month
  Knowledge of 60 nurse managers as assessed using a binary scale (0= No, 1= Yes). Change in nurse managers' knowledge level in one month
Nursing polarity case study situations to assess first-line nurse manager's ability to differentiate between problems to solve and polarities to manage | one month
  Polarity skills of 60 first-line nurse managers as assessed using the dichotomous scale (0= No and 1 = yes)
Questionnaire to measure creativity behavior of first-line nurse managers | one month
  The level of thinking and the ability of nurse managers to produce creative ideas for managing polarities as assessed by a five- Likert scale from 1= never to 5= very often
questionnaire to measure intrinsic work motivation among first-line nurse managers | one month
  intrinsic work motivation among first-line nurse managers as assessed using a five Likert scale (1= strongly disagree, 5= strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Nagah Abd El-Fattah Mohamed Aly, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University, Egypt; Wael M. Lotfy, Ph.D, Study Director — Faculty of Nursing, Matrouh University, Egypt; Safaa M. El-Shanawany, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Maha Ghanem, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Faculty of Nursing, Matrouh University, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No